CLINICAL TRIAL: NCT02882334
Title: Effectiveness Study of Finger Individuation Training by Finger Force Manipulandum (FFM) Compared to Conventional Rehabilitation for Patients With Writer's Cramp
Brief Title: Finger Individuation Training With a Training Device Versus Conventional Rehabilitation for Writer's Cramp
Acronym: FIDEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficultés d'inclure, les patients sont rares
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Foundation Jacques and Gloria Gossweiler (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SSA_2016_15
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Dystonic Disorders
Keywords: Focal Dystonia; Writer's cramp
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Finger individuation training (Experimental): Finger Force Manipulandum
  Interventions: Device: Finger Force Manipulandum
- control (Active Comparator): conventional physiotherapy
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Finger Force Manipulandum
  Arms: Finger individuation training
Other: Conventional physiotherapy
  Arms: control

SUMMARY:
Writer's cramp (WC) is a focal dystonia characterized by abnormal movements and postures during writing. Limited finger independence during writing manifests as difficulty suppressing unwanted activations of neighbouring non task-relevant fingers. WC patients also have difficulty in fine control of grip force. However, some previous studies indicate positive effects of individual finger movement training in WC although these studies lacked enhanced visual feedback of activations in 'stationary' fingers. The investigators have recently developed the Finger Force Manipulandum which quantifies the forces applied by the fingers in different tasks. This method is sensitive for detection and quantification of small unwanted contractions in non-active ('stationary') fingers. Forces in 'stationary' fingers can be displayed on-line providing enhanced feedback on independence of finger movements. The aim of this study is to test the effectiveness of finger individuation training using the FFM to improve symptoms in WC patients.

ELIGIBILITY:
Inclusion Criteria:

* writer's cramp (diagnostic confirmed by a neurologist specialized in movement disorders
* handwriting speed < 140 letters per minute
* simple or complex writer's cramp
* scholarship in French language
* absence of treatment by botulinum neurotoxin, or last injection > 3 months
* age > 18 and < 71 years
* informed consent
* medical insurance coverage

Exclusion Criteria:

* writer's cramp with no impact on writing
* writing tremor
* other neurological disease with effect on writing
* pain or traumatism of the limb used for writing, requiring medical or surgical treatment in the last preceding months
* participation in another research with a potential impact on evaluation criteria
* pregnant or breast feeding patient
* patient under judiciary protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
change in writing speed after rehabilitation | Change from baseline writing speed at week 8
  number of letters correctly copied in 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre BLETON, PhD, Study Chair — Fondation OPH A de Rothschild; Pavel Lindberg, PhD, Study Director — Centre de Psychiatrie et Neurosciences, Inserm U894; Sophie SANGLA, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France